CLINICAL TRIAL: NCT03636607
Title: Diagnostic Significance of Single Center, Open and Prospective Evaluation of <Sup>18<Sup>F-FDG PET/CT Dynamic Imaging and Genomic Sequencing in Detecting Metastatic Lesions of Primary Hepatocellular Carcinoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participents enrolled
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hongjun Jin, Principal Investigator, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ZDWY.FZYX.001
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Positron-Emission Tomography; Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-metastatic group (Experimental): PET/CT dynamic scan,needle biopsy and gene detection
  Interventions: Diagnostic Test: PET/CT dynamic scan
- Metastatic group (Experimental): PET/CT dynamic scan,needle biopsy and gene detection
  Interventions: Diagnostic Test: PET/CT dynamic scan

INTERVENTIONS:
Diagnostic Test: PET/CT dynamic scan — The purpose of this study is to carry out 18F-FDG PET/CT dynamic scans and biopsy of primary or primary and metastatic lesions in newly diagnosed patients with primary liver cancer, and to compare imaging findings, genomics, and pathology at the same time. The intrinsic relationship between tissue characteristics and the diagnostic value of 18F-FDG PET/CT dynamic imaging in primary liver cancer metastases are discussed.
  Other Names: Needle biopasy; Geen detection

SUMMARY:
The aim of this study is to make up for this gap by performing a dynamic scan of 18F-FDG PET/CT on newly diagnosed patients with liver cancer. The lesions and/or metastases are performed for biopsy. Pathological and genomic studies are performed. The differences between tumor images and tissues are compared at the same time. 18F-FDG PET/CT dynamic imaging is explored in primary liver cancer metastases for the diagnostic value.

DETAILED DESCRIPTION:
Hepatic malignancies have a high incidence rate and can be classified into primary liver cancer and metastatic liver cancer according to their sources. There are three main types of primary liver cancer: hepatocellular carcinoma (HCC), cholangiocellular carcinoma (CCC), and mixed hepatocellular carcinoma (both hepatocytes and cholangiolar cells). In recent years, the incidence and mortality of liver cancer have continued to rise. It has high incidence in Southeast Asia and Africa, and the number of liver cancer patients in China accounts for 55% of the world. However, the onset of liver cancer is occult; the degree of malignancy is high, and the progress rate is fast. Most patients have reached late stage or distant metastases when diagnosed. Imaging examination is an important method for the diagnosis and monitoring of liver cancer. The routine imaging examination mainly observed the morphological characteristics and blood supply changes of the liver lesions. The detection rates of CT and MRI for liver cancer can reach 81-89% and 50-80%, respectively. However, these imaging studies have limitations and are vulnerable to local anatomical locations and cannot be used to assess systemic tumor invasion and biological characteristics. Positron emission tomography (PET) is a molecular-level imaging technique that utilizes relatively specific tracers for qualitative and quantitative imaging. The good spatial and density resolutions of computed tomography (X-ray computed tomography, CT) play an important role in the localization and qualitative diagnosis of HCC. 18F-FDG PET/CT can provide functional imaging from the point of view of molecular biology. It not only can understand the tumor invasion of the whole body, but also has become an important means for qualitative diagnosis, staging, prognosis and therapeutic evaluation of tumors.

As a new imaging technology, 18F-FDG PET/CT plays an increasingly important role in the diagnosis of primary liver cancer. 18F-FDG PET/CT reflects the glycometabolism of tumor tissues. The diagnosis of benign and malignant tumors is based on the difference in glucose metabolism between tumor cells and normal tissues. 18F-FDG is an isomer of glucose and is involved in the glucose metabolism process. Since it is deoxygenated, it cannot generate diphosphate hexose, and it cannot participate in the next step of metabolism but remains in the cell. In the tumor cells, due to the high expression of glucose transporter mRNA, the glucose transporters Glut-1 and Glut-3 levels are increased; the expression of hexokinase is increased; the level of glucose-6-phosphatase is down-regulated and other common factors make the tumor cells' 18F-FDG uptake increased.

Previous researchers have found 18F-FDG PET/CT unsatisfactory in the diagnosis of HCC, especially for the diagnosis of HCC with well-differentiated tissue. The researchers also indicates that 18F-FDG PET/CT is not superior to traditional MRI and CT in the diagnosis of liver cancer. Combined with the current relevant research, it can be roughly stated that the positive rate of liver cancer using 18F-FDG PET/CT in diagnosing different grades of tissue differentiation is only about 50-70%. There appears to be a high uptake of FDG in poorly differentiated HCC. However, there is no such obvious phenomenon in HCC with medium or well-differentiated tissue. The PET/CT scans reported in all these documents are based on conventional static scans, i.e. the image data is based on a static take-up image of the tracer in tissue obtained at a fixed time point after the injection of 18F-FDG. To improve, the investigators propose to use dynamic data scanning, which captures the dynamic data of whole body tissues collected from the moment of injecting 18F-FDG to an hour. Dynamic scans can provide information on the dynamic changes in tracer metabolism and distribution in tissues over time, so they provide a richer metabolic and distributional pattern of tumor foci and metastases than static scans. However, the current domestic and international research on 18F-FDG PET/CT dynamic scan in the metastasis of hepatocellular carcinoma is very rare. Therefore, the aim of this study is to make up for this gap by performing a dynamic scan of 18F-FDG PET/CT on newly diagnosed patients with liver cancer. The lesions and/or metastases are performed for biopsy. Pathological and genomic studies are performed. The differences between tumor images and tissues are compared at the same time. 18F-FDG PET/CT dynamic imaging is explored in primary liver cancer metastases for the diagnostic value.

ELIGIBILITY:
Inclusion Criteria:

* Accurately diagnosing primary liver cancer according to pathological diagnostic criteria or clinical diagnostic criteria.
* Tumor volume (> 1 cm) displayed by enhanced CT or MRI or liver mass confirmed by arteriography .
* For patients considering distant metastases, trunk metastases need to be confirmed by CT examination. Bone metastases need to be confirmed by whole-body bone scan. Brain metastases need to be confirmed with characteristic metastatic tumors by MRI.
* The age is more than 18 years old and less than 65 years old. There is no gender restriction.
* Untreated patients who have not received surgery, interventional therapy, chemotherapy, biotherapy, and radiation therapy.
* Physical condition score ECOG: 0-2; no major organ dysfunction; oxygen partial pressure ≥ 10.64kPa; white blood cell count≥ 4 × 109/L; hemoglobin ≥ 9.5g/dL; neutrophil absolute count ≥ 1.5 × 109 / L; platelet count ≥ 100 × 109 / L; total bilirubin ≤ 1.5 times of the upper limit of normal value; creatinine ≤ 1.25 times of the upper limit of normal value; and creatinine clearance ≥ 60ml / min.
* Be able to obtain complete follow-up information, understand the situation of this study and sign informed consent.

Exclusion Criteria:

* Poorly controlled diabetics (fasting blood glucose levels > 200 mg/dL).
* In addition to four types of malignant tumors that can be treated with radical resection, such as cervical cancer in situ, basal or squamous cell skin cancer, (breast) ductal carcinoma in situ, and organ localized prostate cancer, suffering from any other malignant tumors within 5 years.
* Breastfeeding and/or pregnant women.
* Patients with severe bleeding tendencies (prothrombin time less than 50%, cannot be corrected by treatment with vitamin K, etc.).
* Recent severe hemoptysis, severe cough, dyspnea or patients are not able to cooperate.
* People with severe emphysema, pulmonary congestion, and pulmonary heart disease.
* Researchers believe that the subject may not be able to complete this study or may not be able to comply with the requirements of this study (for management reasons or other reasons).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Calculating the overall diagnostic sensitivity and specificity and ROC | 60 minutes
  For each patient enrolled in the study, a two-chamber four-parameter model (2TCM) and a Patlak two-parameter model are established using 18F-FDG PET/CT dynamic scans. Summarizing these dynamic model parameters for all enrolled patients separately calculates the overall diagnostic sensitivity and specificity. Calculate ROC based on sensitivity and specificity.

SECONDARY OUTCOMES:
Calculating the overall diagnostic sensitivity and specificity and summarizing the intrinsic correlations | 60 minutes
  Summarize the genetic testing of all enrolled patients and radiomic indicators to calculate the overall diagnostic sensitivity and specificity. At the same time, the intrinsic correlations between genomics, gene detection and histopathology are summarized.

CONTACTS AND LOCATIONS:
Locations (1):
- Hongjun Jin, Zhuhai, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Undecided